CLINICAL TRIAL: NCT01985776
Title: Effects of Exercise Intervention in Patients With Low Back Pain Due to Spondylolytic Spondylolisthesis
Brief Title: Effects of Exercise Intervention in Patients With Spondylolisthesis Related LBP
Acronym: EXER-SPO-TNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: S2P, Science to Practice, Ltd. (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UP-FVZ-ExerciseSpondylolisth
Record Dates: First submitted 2013-10-30; First posted 2013-11-15 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Low Back Pain; Spondylolisthesis
Keywords: Exercise; Electric Stimulation
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise intervention (Active Comparator): Patients will functional stabilisation exercise for the trunk.
  Interventions: Procedure: Exercise intervention
- Exercise and e-stim (Active Comparator): Patients will receive exercise intervention and electrical stimulation simultaneously.
  Interventions: Procedure: Exercise and e-stim
- Patients control (No Intervention): Patients will not receive any treatment but could use compression belt as per usual.
- Healthy control (No Intervention): Healthy asymptomatic participants who will not receive any treatment.

INTERVENTIONS:
Procedure: Exercise intervention — Functional stabilisation exercise for the trunk.
  Arms: Exercise intervention
Procedure: Exercise and e-stim — Functional stabilisation exercise for the trunk and electrical stimulation at the same time.
  Arms: Exercise and e-stim

SUMMARY:
The first purpose of this study is to define parameters of the trunk neuromuscular functions that are pathologically altered in patients with low back pain due to spondylolytic spondylolisthesis. The second and also the main purpose of the study is to examine the effects of exercise intervention on patients with low back pain due to spondylolytic spondylolisthesis. Our overall hypothesis is that specific exercise intervention will improve neuromuscular functions of the trunk in patients with low back pain due to spondylolytic spondylolisthesis.

DETAILED DESCRIPTION:
Low back pain is known to affect a considerable portion (> 75%) of the society, causing enormous financial burden for the healthcare systems.

Exercise interventions incorporated into low back pain patients rehabilitation protocols are known as successful treatment strategies, but ore often focused on strength training and not on functional stabilization. Spondylolytic spondylolisthesis is one of the most known types of spine instabilities. To date, no studies examined the effects of exercise intervention on patients with low back pain due to spondylolytic spondylolisthesis. Research will be carried out as a cross-sectional study, where patients with spondylolytic spondylolisthesis will be randomly arranged in one controlled and two experimental groups. For the forth group healthy asymptomatic participants will be recruited.

Exercise intervention will last 12 weeks with a frequency of three times a week and duration of 60 minutes per training unit. Exercise intervention will include congregated set of trunk stabilisation exercises, starting with simple isometric tasks. Dynamic and more complex movements will be added progressively to achieve whole body tasks involving fast and sudden movements.

Neuromuscular functions of the trunk will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain presence for at least three months.
* Age between 20 and 60 years.
* Isthmic Spondylolisthesis (1st and 2nd level according to Meyerding) at L5/S1 and L4/L5.
* Body mass index below 30.
* without neurological pathological conditions.

Exclusion Criteria:

* Intermittent claudication pain.
* History of operational treatment of the lumbar spine.
* Traumatic, oncological, infectional pathology of the spine
* Degenerative stenosis of the lumbar spinal canal.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in measures of neuromuscular functions of the trunk | Change from baseline values at 9 weeks
  Set of tests that objectively evaluate the neuromuscular functions of the trunk.
  * Ability to reposition the trunk position during forward bent
  * Maximal voluntary contraction during trunk flexion, extension and lateral flexion
  * Muscle endurance during isometric trunk extension.
  * Trunk's muscles activation during sudden loading and fast arm movement
  * Single leg stance
  * Leg symmetry during squat
  * Hip and spine flexibility

SECONDARY OUTCOMES:
Changes in Oswestry questionnaire score | Change from baseline values at 9 weeks
  Oswestry Low Back Pain Questionnaire commolny used by clinicians and researchers to quantify disability for low back pain.
Change in Posture parameters | Change from baseline values at 9 weeks
  Angular and linear posture measures in frontal and sagittal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Sarabon, PhD, Principal Investigator — University of Primorska
Locations (4):
- Slovenia (4):
  - Orthopaedic Hospital Valdoltra, Ankaran
  - University of Primorska, Science and Research Centre of Koper, Institute for Kinesiology Research, Koper
  - University Medical Centre Ljubljana, Ljubljana
  - University Medical Centre Maribor, Maribor